CLINICAL TRIAL: NCT06675890
Title: Correlation of Serum Homocysteine Levels With Various Types of Coronary Artery Disease (CAD) and In-hospital Mortality
Brief Title: Homocysteine and Coronary Artery Disease
Status: Completed | Type: Observational
Sponsor: Shaqra University (Other)
Responsible Party: Principal Investigator, Himayat Ullah, Assistant Professor/Dr, Shaqra University
Other Study IDs: 599/HEC/B&PSE/2021
Record Dates: First submitted 2024-11-01; First posted 2024-11-05 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Coronary Arterial Disease (CAD)
Keywords: Coronary Artery Disease; Serum Homocysteine; In-hospital Mortality
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients having coronary arterial disease.: patients with different types of coronary arterial disease and their homocysteine levels.
  Interventions: Diagnostic Test: serum homocysteine

INTERVENTIONS:
Diagnostic Test: serum homocysteine — serum homocysteine is associated with atherosclerosis and vascular diseases.

SUMMARY:
This study is aimed at correlating serum homocysteine level with coronary artery disease (CAD) and related in-hospital mortality. A cross section of patients from age 18 years and above will be studied for homocysteine level and analyzed for the above mentioned correlation. The study was approved by hospital ethical review board as mentioned. An informed written consent was obtained before the patients' recruitment.

DETAILED DESCRIPTION:
This study explores the correlation between serum homocysteine levels, coronary artery disease (CAD), and in-hospital mortality, addressing the need to understand homocysteine's role as a potential marker for CAD severity and mortality risk. Homocysteine is an amino acid linked to vascular inflammation and endothelial damage, both critical factors in cardiovascular pathology. Elevated homocysteine levels, often stemming from genetic predispositions or lifestyle factors like poor diet and smoking, are associated with endothelial dysfunction, plaque formation, and thrombotic complications, all of which are common in CAD patients. Thus, investigating this correlation is essential, as it may reveal whether homocysteine levels can reliably predict CAD outcomes or mortality risk in hospitalized patients, potentially impacting future diagnostic and therapeutic protocols.

Study Design and Methodology The study adopts a cross-sectional design to assess patients aged 18 years and older, utilizing serum homocysteine level testing and correlational analyses with CAD severity and mortality outcomes. A cross-sectional study is particularly suitable for identifying associations and trends within a specific population at a single point in time, making it advantageous for examining homocysteine's role in CAD. The study captures a broad spectrum of CAD presentations and risk profiles by including adult patients from various backgrounds. This allows for a more comprehensive analysis of homocysteine levels in various CAD contexts, from mild cases to severe in-hospital mortalities.

The study's inclusion of patients above 18 years ensures a diverse age demographic, crucial for understanding homocysteine's role in different age-related presentations of CAD. It allows for subgroup analyses to observe how age may influence homocysteine's effects on CAD progression or outcomes, as younger and older patients may exhibit differing metabolic and vascular responses. Homocysteine levels are influenced by various physiological, lifestyle, and genetic factors, which can vary across age groups. Observing these distinctions can add depth to our understanding of CAD in relation to homocysteine.

Ethical Considerations and Consent The ethical framework of this study is paramount, especially in a hospital setting with vulnerable patients. Approval from the hospital's ethical review board underpins the study's commitment to ethical standards, ensuring that the research adheres to principles such as patient confidentiality, respect, and transparency. Ethical board approval also reflects adherence to institutional standards for patient welfare and safety. Participants were informed of the study's objectives, procedures, and potential implications, allowing them to make an informed decision about participation. Written informed consent ensures patients voluntarily agree to partake, providing them with an understanding of their participation and rights as subjects.

Informed consent also means participants understand that their serum homocysteine levels will be evaluated alongside their CAD diagnosis and outcomes, making them aware of potential benefits and risks. The consent process ensures voluntary participation, empowering patients and fostering trust. As part of ethical considerations, the study includes provisions for confidentiality, ensuring patients' data is used only for research purposes and stored securely to protect personal health information.

Serum Homocysteine as a Potential Biomarker Homocysteine's significance as a potential biomarker stems from its biochemical interactions within the body. Homocysteine is an intermediary in the metabolic pathway of methionine, a sulfur-containing amino acid obtained from dietary protein. Elevated homocysteine levels, known as hyperhomocysteinemia, result from disruptions in this pathway due to genetic factors, lifestyle habits, or inadequate intake of essential vitamins like B6, B12, and folate. Elevated homocysteine levels are linked to endothelial cell injury, oxidative stress, and the formation of atherosclerotic plaques, contributing to CAD pathogenesis.

In this study, measuring serum homocysteine levels in patients with CAD could reveal correlations between elevated homocysteine and disease severity and short-term mortality. Hyperhomocysteinemia has been associated with several pathophysiological mechanisms, such as pro-inflammatory and pro-coagulant states that favor plaque instability and thrombosis. Therefore, if serum homocysteine levels consistently correlate with severe CAD or increased mortality, it could serve as a practical biomarker for identifying high-risk CAD patients in clinical settings. Homocysteine level measurement is relatively accessible and cost-effective, offering a practical advantage for early risk assessment and monitoring.

Statistical Analysis and Hypothesis Testing The study employs statistical tests such as ANOVA, Kruskal-Wallis, Tukey's post hoc, Pearson correlation, and binary regression analysis to analyze the relationship between serum homocysteine levels and CAD severity. These methods allow researchers to assess whether homocysteine levels significantly differ across types of CAD and whether they predict in-hospital mortality.

1. ANOVA and Kruskal-Wallis Tests: These tests assess variations in homocysteine levels across different CAD categories. The one-way ANOVA, complemented by the non-parametric Kruskal-Wallis test, helps confirm the robustness of findings, ensuring that homocysteine's relationship with CAD holds true even in samples with non-normal distributions.
2. Tukey's Post Hoc Test: Following ANOVA, Tukey's post hoc test identifies specific group differences, pinpointing which types of CAD show the strongest association with elevated homocysteine.
3. Pearson Correlation: This correlation measures the strength and direction of the relationship between homocysteine levels and CAD severity. Initial results suggest a moderate positive correlation. A correlation of 0.4, as noted in the abstract, indicates a moderate link, suggesting that higher homocysteine may be moderately predictive of CAD presence and severity.
4. Binary Regression Analysis: To explore homocysteine as a predictor of in-hospital mortality, binary regression analysis estimates the mortality risk increase with each unit increase in homocysteine. This analysis revealed that each 1 µmol/L rise in homocysteine is associated with a 10.5% increase in mortality risk, highlighting its potential as a prognostic marker.

Implications and Potential Applications If the findings support serum homocysteine as a reliable marker for CAD and mortality, this could influence CAD risk assessment practices. Homocysteine screening could become part of routine CAD evaluation, helping identify high-risk patients who may benefit from more intensive monitoring or early interventions. Elevated homocysteine could prompt lifestyle or pharmacological interventions to lower levels, potentially improving cardiovascular outcomes. For example, patients with high homocysteine might benefit from B-vitamin supplementation to lower levels and mitigate CAD risk, though further studies are required to confirm clinical benefits.

Furthermore, identifying homocysteine's role in CAD could open avenues for tailored treatments. In patients with elevated homocysteine, therapies targeting endothelial protection, anti-inflammatory strategies, or specific dietary recommendations may offer added benefits. If validated in larger studies, homocysteine could emerge as an essential biomarker in CAD prognosis, offering insights that could personalize treatment plans based on biochemical markers beyond traditional risk factors.

Limitations and Future Directions The study's cross-sectional design, while valuable for identifying associations, limits the ability to infer causality between homocysteine and CAD. Longitudinal studies would be necessary to establish whether elevated homocysteine levels directly contribute to CAD progression or if they are secondary to underlying cardiovascular pathology. Another limitation is the reliance on single homocysteine measurements, which may fluctuate due to dietary and lifestyle factors. Repeated measurements could provide more accurate insights into homocysteine's relationship with CAD and mortality.

Future studies could expand on this research by examining larger and more diverse populations, enhancing the findings' generalizability. Additionally, exploring genetic factors that influence homocysteine metabolism, such as polymorphisms in methylenetetrahydrofolate reductase (MTHFR), could reveal whether specific genetic profiles predispose individuals to higher CAD risk. Investigating interactions between homocysteine and other biomarkers, like CRP or fibrinogen, may also offer a multi-dimensional understanding of CAD risk.

Conclusion This study is a significant step in understanding serum homocysteine's role in CAD and its potential as a mortality predictor in hospitalized patients. By evaluating homocysteine's relationship with CAD types and in-hospital mortality, the study adds to the growing body of evidence on homocysteine as a marker for cardiovascular risk. If validated, serum homocysteine measurement could be an accessible tool for assessing CAD severity and tailoring treatment strategies, ultimately contributing to improved cardiovascular care outcomes.

ELIGIBILITY:
Inclusion Criteria:

• Coronary artery disease patients from age 25 years to 80 years.

Exclusion Criteria:

* Grade 4 chronic kidney disease patients
* Chronic liver disease patients
* Pregnant and lactating females
* Patients on vitamin supplements
* Patients with genetic homocysteine abnormalities

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of all ethnicities and both genders from 25 to 80 years with coronary artery disease.
Sampling Method: Non-Probability Sample
Enrollment: 381 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Homocysteine levels and its correlation with the type of coronary artery disease. | 2 years
  Higher homocysteine levels in ST segment myocardial infarction (STEMI) and non ST segment myocardial infarction (NSTEMI) as compared to Angina.

SECONDARY OUTCOMES:
Risk factors for coronary artery disease | 2 years
  Other biochemical risk factors of coronary artery disease, like serum fibrinogen, hsCRP, Serum cholesterol levels

CONTACTS AND LOCATIONS:
Overall Officials: Himayat Ullah, FCPS, Principal Investigator — Shaqra University
Locations (1):
- Hayatabad Medical Complex, Peshawar, KPK, Pakistan

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared due to confidentiality.

REFERENCES:
- [Background] Hankey GJ, Eikelboom JW. Homocysteine and vascular disease. Lancet. 1999 Jul 31;354(9176):407-13. doi: 10.1016/S0140-6736(98)11058-9. PMID 10437885
- [Background] Ridker PM, Hennekens CH, Buring JE, Rifai N. C-reactive protein and other markers of inflammation in the prediction of cardiovascular disease in women. N Engl J Med. 2000 Mar 23;342(12):836-43. doi: 10.1056/NEJM200003233421202. PMID 10733371
- [Background] Roth GA, Mensah GA, Johnson CO, Addolorato G, Ammirati E, Baddour LM, Barengo NC, Beaton AZ, Benjamin EJ, Benziger CP, Bonny A, Brauer M, Brodmann M, Cahill TJ, Carapetis J, Catapano AL, Chugh SS, Cooper LT, Coresh J, Criqui M, DeCleene N, Eagle KA, Emmons-Bell S, Feigin VL, Fernandez-Sola J, Fowkes G, Gakidou E, Grundy SM, He FJ, Howard G, Hu F, Inker L, Karthikeyan G, Kassebaum N, Koroshetz W, Lavie C, Lloyd-Jones D, Lu HS, Mirijello A, Temesgen AM, Mokdad A, Moran AE, Muntner P, Narula J, Neal B, Ntsekhe M, Moraes de Oliveira G, Otto C, Owolabi M, Pratt M, Rajagopalan S, Reitsma M, Ribeiro ALP, Rigotti N, Rodgers A, Sable C, Shakil S, Sliwa-Hahnle K, Stark B, Sundstrom J, Timpel P, Tleyjeh IM, Valgimigli M, Vos T, Whelton PK, Yacoub M, Zuhlke L, Murray C, Fuster V; GBD-NHLBI-JACC Global Burden of Cardiovascular Diseases Writing Group. Global Burden of Cardiovascular Diseases and Risk Factors, 1990-2019: Update From the GBD 2019 Study. J Am Coll Cardiol. 2020 Dec 22;76(25):2982-3021. doi: 10.1016/j.jacc.2020.11.010. PMID 33309175
- [Background] Wong ND. Epidemiological studies of CHD and the evolution of preventive cardiology. Nat Rev Cardiol. 2014 May;11(5):276-89. doi: 10.1038/nrcardio.2014.26. Epub 2014 Mar 25. PMID 24663092
- [Background] Khan MA, Hashim MJ, Mustafa H, Baniyas MY, Al Suwaidi SKBM, AlKatheeri R, Alblooshi FMK, Almatrooshi MEAH, Alzaabi MEH, Al Darmaki RS, Lootah SNAH. Global Epidemiology of Ischemic Heart Disease: Results from the Global Burden of Disease Study. Cureus. 2020 Jul 23;12(7):e9349. doi: 10.7759/cureus.9349. PMID 32742886